CLINICAL TRIAL: NCT00005112
Title: Growth Hormone Use in Cystic Fibrosis - a Multicenter Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Genentech, Inc. (Industry)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: NCRR-M01RR02558-0111; M01RR002558 (NIH); NCT00000109 (obsolete NCT alias)
Record Dates: First submitted 2000-04-15; First posted 2000-04-17 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

INTERVENTIONS:
Drug: Human recombinant growth hormone

SUMMARY:
Cystic Fibrosis (CF) is the most common lethal genetic disorder in America. Previous studies by our group and others have shown that human recombinant growth hormone (GH) improves height velocity, weight velocity, lean body mass (LBM) and pulmonary function. These positive results have prompted us to ask further questions regarding GH use in CF including: a) Do patients with better baseline body weight and pulmonary function derive more benefit from treatment than those with worse weight and pulmonary function?, b) Does GH use improve the patient's quality of life?, c) Once GH is discontinued, are the positive effects sustained? We hypothesize that GH treatment in CF patients will improve their clinical status and their quality of life. We further hypothesize that these effects will be present regardless of baseline body weight or pulmonary function, and that positive outcome will be sustained for at least one year after GH treatment is discontinued. To test our hypothesis, we will recruit 40 prepubertal children from five CF centers across the United States (8 per center). Patients will be randomly assigned to receive treatment with GH (0.3mg/kg/wk) during either the first or the second year. All subjects will be seen every three months. We will evaluate the following parameters every three months: 1) height, height velocity and Z-score, 2) body weight and weight velocity. Every six months we will measure: 1) lean body mass utilizing DEXA, 2) pulmonary function, including measurement of respiratory muscle strength (peak inspiratory and peak expiratory pressure), 3) quality of life (QOL), quantitated from QOL forms specific for CF ("The Cystic Fibrosis Questionnaire"). After one year of study, subjects will "cross-over" to the other treatment arm. This 24 month study will allow us to statistically compare outcome measures in 20 treated and 20 nontreated subjects from multiple centers, and will allow us to assess sustained effect in the 20 subjects who receive GH during the first year, by comparing their results to results obtained during the year post treatment.

ELIGIBILITY:
Inclusion Criteria:

* CF patients ages 5-12 who are less than the 25th percentile for age and sex normal values for height and/or weight

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child

CONTACTS AND LOCATIONS:
Overall Officials: Dana Hardin, M.D., Principal Investigator
Locations (2):
- United States (2):
  - University of Texas Medical School, Houston, Texas
  - University of Utah, Dept of Pediatric Endocrinology, Salt Lake City, Utah